CLINICAL TRIAL: NCT05925244
Title: A Preliminary Study on the Effect of Loaded and Unloaded Exercise on Anabolic and Turnover Activity of Articular Cartilage in Healthy Young Adults
Brief Title: The Anabolic and Catabolic Effect of Loaded and Unloaded Exercise on Articular Cartilage Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HS22322
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: articular cartilage; walking exercise; sCOMP; PIIANP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Experimental): The control condition did 30 minutes of walking exercise with their own body mass.
  Interventions: Other: Control Condition
- +12% Body Mass (Experimental): The +12% body mass condition did 30 minutes of walking exercise wearing a weighted vest with +12% of their body mass applied.
  Interventions: Other: +12% Body Mass
- -12% Body Mass (Experimental): The -12% body mass condition did 30 minutes of walking exercise using a lower body positive pressure treadmill with -12% of their body mass applied.
  Interventions: Other: -12% Body Mass

INTERVENTIONS:
Other: Control Condition — Control (no alteration to body mass).
  Arms: Control
Other: +12% Body Mass — Loaded walking exercise (12% increase in body mass using a weighted vest).
  Arms: +12% Body Mass
Other: -12% Body Mass — Unloaded walking exercise (12% decrease in body mass using lower body positive pressure).
  Arms: -12% Body Mass

SUMMARY:
The serum concentration of cartilage oligomeric matrix protein (sCOMP) has been considered a mechano-sensitive biomarker of articular cartilage turnover, and N-propeptide of type II collagen (PIIANP) is a proposed biomarker of type II collagen synthesis. Few studies have investigated both the anabolic and turnover response of articular cartilage as a result of acute changes in body weight mass during exercise. Using a repeated measures cross-over design, fifteen healthy adults (age 18-30 years) performed three, 30-minute bouts of treadmill walking exercise under 3 loading conditions: (1) control (no alteration to body mass); (2) loaded (12% increase in body mass using a weighted vest); and (3) unloaded (12% decrease in body mass using lower body positive pressure). Venous blood was collected before, immediately after, and 15 and 30 minutes after exercise to investigate cartilage turnover (sCOMP) and anabolism (PIIANP).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18-30 years old

Exclusion Criteria:

* Traumatic injury to the lower extremity in the past year
* Hip, knee, or ankle surgery
* Radiographic evidence of joint degeneration
* Cardiovascular disease
* Ankylosing spondylitis
* Psoriatic arthritis
* Chronic reactive arthritis
* Renal problems requiring peritoneal dialysis or hemodialysis
* Not currently using any prescription or non-prescription medications and/or nutritional supplements

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Serum cartilage oligomeric matrix protein (sCOMP) | sCOMP was measured at baseline, immediately post, and 15- and 30-minutes post exercise.
  The systemic blood serum concentration of sCOMP was evaluated in all participants under the 3 conditions in a crossover trial.
N-propeptide of type II collagen (PIIANP) | PIIANP was measured at baseline, immediately post, and 15- and 30-minutes post exercise.
  The systemic blood serum concentration of PIIANP was evaluated in all participants under the 3 conditions in a crossover trial.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cornish, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
The data will not be available to other researchers as we do not have ethical approval to do so.

REFERENCES:
- [Derived] de Vasconcelos BM, Peeler JD, Scribbans T, Cornish SM. A preliminary study on the effect of loaded and unloaded exercise on N-propeptide of type II collagen and serum cartilage oligomeric matrix protein activity of articular cartilage in healthy young adults. Appl Physiol Nutr Metab. 2023 Dec 1;48(12):954-961. doi: 10.1139/apnm-2023-0124. Epub 2023 Aug 9. PMID 37556859